CLINICAL TRIAL: NCT04014855
Title: The Effect of Lactoferrin Versus Iron Supplement in Treating Iron Deficiency Anemia and Helping Weight Loss in Obese School Age Children
Brief Title: Lactoferrin Versus Iron Supplement in Irondeficiency Anemia and Weight Loss in Obese Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Marian girgis, lecturer of paediatrics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 271182
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity | interventions — Iron-Dextran Complex; Lactoferrin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- obese children 1 (Active Comparator): iron supplementation
  Interventions: Drug: Iron Supplement
- obese children 2 (Active Comparator): lactoferrin supplementation
  Interventions: Drug: Iron Supplement

INTERVENTIONS:
Drug: Iron Supplement — in iron deficiency anemia
  Other Names: lactoferrin

SUMMARY:
The effect of lactoferrin versus iron supplement in treating iron deficiency anemia and helping weight loss in obese school age children

DETAILED DESCRIPTION:
Comparing iron versus lactoferrin as regard iron defiency anemia and weight loss in obese children

ELIGIBILITY:
Inclusion Criteria:

* 1. children age will be between 6 -12 years old. 2. Presence of iron deficiency anemia, it will be diagnosed by

  * CBC >> Hemoglobin level concentration below 11.5 g/dl.
  * level of serum iron is below 30 µmol/l,
  * level of ferritin is below 15 µg/dl
  * Total iron binding capacity is more 480 µg/dlL. 3. children should be stable and free from chronic disease. 4. Body Mass index (BMI) should be ≥the 95th percentile for children and teens of the same age and sex.

    5. there is not history of iron supplements in the 3 months before treatment.

Exclusion Criteria:

1. Father/mother refuses to participate in the study.
2. Hospitalized patient.
3. Non-anemic patient.
4. Patients receiving iron supplements 3 months before enrollment.
5. Patients with chronic diseases.
6. personal or family history of allergy to cow's milk or infant formula, eczema, moderate-to-severe allergic rhinitis or asthma, or milk intolerance.
7. severe anemia as Hemoglobin level concentration below 7 g/dl.

Exclusion Criteria:

-

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
iron deficiency anemia | 3 months
  CBC and iron profile

SECONDARY OUTCOMES:
weight | 3 months
  Weight and body copmositiin

CONTACTS AND LOCATIONS:
Overall Officials: Marian GR Abdelsayed, Principal Investigator — Ain Shams University
Locations (1):
- Marian Girgis Rizk Abdelsayed, Cairo, Non-US/Non-Canadian, Egypt

IPD SHARING:
Plan to Share IPD: No